CLINICAL TRIAL: NCT05226832
Title: Intradetrusor Triamcinolone Injection in the Management of Interstitial Cystitis/Bladder Pain Syndrome: Pilot Study
Brief Title: Intradetrusor Triamcinolone Injection in the Management of Interstitial Cystitis/Bladder Pain Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-0227
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Injection Group (Experimental)
  Interventions: Procedure: 40mg Triamcinolone Injections in the Bladder

INTERVENTIONS:
Procedure: 40mg Triamcinolone Injections in the Bladder — Patients will undergo a standard of care cystoscopy with non-standard of care solumedrol injections in the clinic. Subjects will have lidocaine jelly instilled into their bladder for 5 minutes prior to injection cystoscopy. Injections will be performed using a 17fr flexible cystoscope in the outpatient setting. There will be 10 intravesical Injections of 1cc of 40mg solumedrol diluted to 10cc with injectable normal saline. The needle will penetrate the bladder at a depth of 2-3mm using a Laborie endoscopic single use needle, about the length of a pencil tip. The patient may experience discomfort with cystoscopy and injections. Any procedure complications will be noted based on the Clavien-Dindo Classification Index, discussed in the safety section. This is estimated to take 30 minutes.

SUMMARY:
This initial pilot project aims to study the use of FDA-approved 40mg triamcinolone injections in the bladder for the management of interstitial cystitis with or without Hunner's lesions. Intradetrusor triamcinolone injections are already the standard of care for IC patients with Hunner's lesions, but its role in management of IC without Hunner's lesions has yet to be determined. Triamcinolone is a long-acting corticosteroid that acts by inhibiting the migration of polymorphonuclear leukocytes, which may contribute to attenuation of inflammation in interstitial cystitis. We will recruit 27 females 18 years of age or older that have been diagnosed with IC/BPS. Patients will undergo a one-time cystoscopy along with the triamcinolone injections for IC management as a part of the research study. Validated questionnaires will be provided before the treatment to quantify symptoms at baseline and after treatment at follow-up visits. Follow up visits will occur in clinic every 4 to 6 weeks, which will continue for a maximum of 1 year. Scores at follow-up visits will be compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet an appropriate diagnosis of IC from NIDDK (National Institute of Diabetes and Digestive and Kidney Diseases)
* Patients must be female
* 18 years or older
* Have an official diagnosis of Interstitial Cystitis/Bladder Pain Syndrome

Exclusion Criteria:

* Patients who do not meet NIDDK inclusion criteria for Interstitial Cystitis as described above will not me enrolled in the study
* The presence of urinary tract or sexually transmitted infection (may be included once existing infection is treated and cleared)
* Pregnant women
* Patients who have the inability to consent on their own behalf
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
O'Leary-Sant Symptom Index; Problem Index; Pain, Urgency, Frequency Symptom Scale | One Year
  Follow-up visits will occur every 4-to-6-weeks post-procedure as part of UTMB's standard of care. Patients will be asked to fill out The O'Leary-Sant Symptom Index and Problem Index and the Pain, Urgency, Frequency Symptom Scale to quantify symptoms, which is not experimental. No other procedures will occur for Visits #3 and onward. Follow-up visits will continue for a maximum of 1 year

IPD SHARING:
Plan to Share IPD: No